CLINICAL TRIAL: NCT07379281
Title: Research Protocol for Evaluating the Efficacy of Neoadjuvant Chemotherapy Drugs for Muscle-Invasive Bladder Cancer Based on Organoid Technology.
Brief Title: Evaluating the Efficacy of Neoadjuvant Chemotherapy Drugs Based on Organoid Technology
Status: Recruiting | Type: Observational
Sponsor: Qilu Hospital of Shandong University (Other)
Collaborators: The Second Hospital of Shandong University (Other); Qianfoshan Hospital (Other); Shandong Provincial Hospital (Other Government); Shandong Province Third hospital (Other); Taian City Central Hospital (Other); Weifang People's Hospital (Other); Binzhou Medical University (Other); The Affiliated Hospital of Qingdao University (Other); Jining First People's Hospital (Other); Liaocheng People's Hospital (Other); Linyi People's Hospital (Other); Yantai Yuhuangding Hospital (Other); Zibo Central Hospital (Other Government); Dezhou Hospital Qilu Hospital of Shandong University (Other); Zaozhuang Municipal Hospital (Other); Qilu Hospital of Shandong University (Qingdao) (Other)
Responsible Party: Sponsor
Other Study IDs: KYLL-202411-011-1
Record Dates: First submitted 2026-01-23; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-12

CONDITIONS: Bladder Cancer
Keywords: Organoid; Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Experimental group: Using tumor organoid drug sensitivity tests to assess the sensitivity of patients' tumor cells to six neoadjuvant chemotherapy drugs, in order to develop a neoadjuvant chemotherapy regimen.
  Interventions: Other: Organoid culture
- Control group: Bladder cancer patients who underwent radical surgery during the same period and received neoadjuvant chemotherapy according to the standard regimen were selected as the control group.

INTERVENTIONS:
Other: Organoid culture — Organoid culture of tumor tissue obtained during patient surgery
  Groups: Experimental group

SUMMARY:
This study, through a clinical controlled trial, compared the one-year, three-year, and five-year overall survival rates between patients receiving a treatment plan guided by organoid drug sensitivity and those receiving conventional empirical treatment. Univariate Kaplan-Meier survival analysis was used to compare the differences in overall survival between the two groups. The study aimed to evaluate the application value of tumor organoid drug sensitivity testing in guiding neoadjuvant chemotherapy for bladder cancer.

DETAILED DESCRIPTION:
1. Research Background (Stating the Rationale and Significance of This Study by Combining Domestic and International Research Status)

   Bladder cancer is a malignant tumor originating from the urothelium of the bladder and ranks first in incidence among urogenital tumors in China. Among these, urothelial carcinoma is the most common, accounting for over 90% of bladder cancer cases [1]. Based on the depth of tumor invasion and prognostic characteristics, bladder cancer is clinically classified into non-muscle-invasive bladder cancer (NMIBC) and muscle-invasive bladder cancer (MIBC). MIBC constitutes approximately 20% of newly diagnosed bladder cancer cases [2-3], but its prognosis is significantly worse than that of NMIBC, with a 5-year overall survival (OS) rate of about 60%-70% [4-5].

   For patients with T2~T4a stage disease without distant metastasis, radical cystectomy (RC) is typically the primary treatment. However, despite undergoing RC and pelvic lymph node dissection, about 50% of patients ultimately experience tumor progression due to disseminated metastasis [2-3]. Therefore, combining systemic therapy with surgery plays a crucial role in reducing tumor progression rates. Cisplatin-based neoadjuvant chemotherapy (NAC) was first evaluated as a potential treatment strategy for MIBC in the 1980s and showed promising efficacy [6]. Subsequent studies have associated NAC-induced downstaging of MIBC with improved survival rates [7-8]. The BA06 30894 trial is the largest NAC study in bladder cancer to date. In this trial, 976 patients received either neoadjuvant cisplatin, methotrexate, and vinblastine (CMV) or no NAC before RC and/or radiotherapy. With a median follow-up of 8 years, the use of neoadjuvant CMV increased the 10-year survival rate from 30% to 36% (HR, 0.84; 95% CI, 0.72-0.99; P = .037) [9-10]. For bladder cancer patients, NAC can maximally eradicate tumor cells, reduce tumor volume, lower clinical stage, thereby increasing the chance of complete surgical resection, and prevent potential tumor dissemination caused by surgical manipulation. Consequently, cisplatin-based NAC has become the standard treatment for eligible MIBC patients according to most international guidelines [11]. Currently, commonly used neoadjuvant chemotherapy agents include [12]: cisplatin, gemcitabine, methotrexate, vinblastine, doxorubicin... However, precisely due to the variety of NAC drugs and differing administration methods, the selection of chemotherapy regimens often relies on physicians' clinical experience or specific research findings, lacking a unified standard, and is characterized by blindness, empiricism, and randomness. Furthermore, some patients exhibit intrinsic resistance to certain chemotherapeutic agents. By the time clinical assessment confirms a patient's insensitivity to the applied drug, severe toxic side effects have already occurred, potentially even leading to multi-drug resistance (MDR), depriving the patient of the opportunity to choose alternative treatments. Therefore, how to evaluate NAC responsiveness, avoid primarily resistant drugs, and directly select highly sensitive agents to achieve individualized chemotherapy has become a hotspot in NAC research.

   The realization of precise cancer treatment largely depends on drug sensitivity testing. Through precise and individualized chemotherapy drug screening tests, the most effective and least toxic treatment plan can be determined for each patient before therapy begins. Proposing a chemotherapy regimen tailored to the individual patient represents a new research direction for achieving precision treatment in bladder cancer and improving chemotherapy response rates. Previously, the more commonly used preclinical models were traditional tumor cell lines and patient-derived xenograft (PDX) models. While tumor cell line culture is simple, it is insufficient to simulate the growth state of tumor cells in the patient's body, and the drugs screened by this system have low clinical application value. Although PDX models can simulate in vivo tumor characteristics and preserve the tumor microenvironment, they have significant limitations, such as relatively low stable engraftment rates, long modeling and evaluation cycles (six months to one year), being time-consuming and labor-intensive, making them difficult to generate and use for high-throughput drug screening [13-16]. Therefore, to develop more personalized treatment and prevention strategies tailored to an individual's unique genetic, environmental, and lifestyle characteristics, minimizing risks and optimizing medical intervention outcomes, it is essential to develop drug sensitivity testing models that can simulate the heterogeneity and complexity of bladder cancer.

   Organoids, specifically Patient-Derived Organoids (PDOs), are three-dimensional organotypic structures formed through the self-assembly of stem cells in vitro. They can differentiate into multiple organ-specific cell types and exhibit cell-cell interactions, cell-extracellular matrix interactions, and spatial organization, thereby recapitulating some key functions and structures of real human organs in vitro while maintaining stable phenotypic and genetic characteristics. Compared to two-dimensional tumor cell lines and PDX models, tumor organoids can be directly cultured from a patient's own tissue. These organoids can effectively replicate key properties of the primary tumor, preserve the pathological morphology and biological mechanisms of the patient's tissue, retain tumor heterogeneity and a more authentic tumor microenvironment, and have the advantage of a short growth cycle [17]. This facilitates their use for sensitivity testing of chemotherapy drugs, molecularly targeted agents, anti-tumor antibodies, etc., in clinical cancer patients, predicting patient response to drugs, and holds potential for assisting clinical treatment decision-making.

   In 2018, a study published in Science reported the use of metastatic gastrointestinal cancer organoids for drug sensitivity testing [18]. This study compared and analyzed the differences in sensitivity to a series of targeted and chemotherapeutic drugs between 21 clinical patients and their corresponding PDOs, demonstrating strong consistency between the two. Compared with the patients' actual therapeutic outcomes, the PDO predictions were robust (sensitivity 100%, specificity 93%, positive predictive value 88%, and negative predictive value 100%). In 2020, Yao Y et al. [19] utilized biopsy tissues from 112 patients with locally advanced rectal cancer to construct 96 rectal cancer organoids. Eighty of these were selected to test their response to chemoradiotherapy, and the results showed that the sensitivity of rectal cancer organoids to chemoradiotherapy was highly consistent with the patients' clinical responses (sensitivity 78%, specificity 92%, accuracy 84%). Subsequently, consistency between PDO drug response and patient clinical response has also been observed in gastric cancer, breast cancer, and other tumors. Yan HHN et al. [20] established a gastric cancer organoid biobank using tumor tissues, adjacent normal tissues, and lymph node metastasis samples from 34 gastric cancer patients. Among them, two cases developed metastasis and received postoperative combination therapy with cisplatin and 5-FU, both showing good responses. Another case received preoperative chemotherapy and showed no response to postoperative capecitabine. Investigating the sensitivity of the PDOs from these three cases to the corresponding compounds revealed that the drug sensitivity of the PDOs was completely consistent with the clinical responses of the respective patients. Guillen KP et al. [21] generated PDX and PDO models from tumor samples of breast cancer patients with endocrine therapy resistance, recurrence, and metastasis, and performed histomorphological, genomic, and drug sensitivity analyses on these samples. The results indicated that both breast cancer PDX and PDO models highly recapitulated the tissue biology and genomics of their source tumors, and their responses to anti-tumor drugs were consistent. In this study, a patient with stage IIA triple-negative breast cancer developed liver metastasis approximately one year after undergoing preoperative chemotherapy and surgery. The researchers conducted in vitro and in vivo drug sensitivity tests on the constructed PDO and PDX models and found that the microtubule inhibitor eribulin had the best therapeutic effect. Based on this finding, the patient was guided to receive eribulin treatment, resulting in complete remission of the liver metastasis lasting nearly 5 months. These studies provide preliminary evidence for the potential of PDOs to guide clinical drug use for cancer patients. Additional research has shown that by comparing the drug response differences between normal organoids and PDOs, highly selective drugs can be identified, which may help reduce toxic side effects in clinical patients. Thus, conducting drug sensitivity testing via PDOs to discover the most suitable drug treatment plan will help improve clinical efficacy for cancer patients, reduce toxic side effects, the risk of drug resistance, and the likelihood of tumor progression, maximizing patient benefit.

   Therefore, leveraging patient-derived bladder cancer organoid models to conduct neoadjuvant chemotherapy drug sensitivity testing for muscle-invasive bladder cancer, establishing a standardized bladder cancer organoid drug sensitivity testing system, and formulating screening criteria for bladder cancer organoid drug sensitivity testing, will enable the selection of optimal neoadjuvant drug combination regimens. This approach can assist in developing novel individualized treatment plans for clinical application and undergo multi-center clinical validation, ultimately achieving true "avatar drug testing."
2. Research Questions and Objectives (Elucidating the Scientific Questions and Research Objectives)

Research Question: This study employs a clinical controlled trial design to compare the one-year, three-year, and five-year overall survival rates between a patient group receiving interventions guided by organoid drug sensitivity testing and a patient group receiving traditional empirical treatment. Univariate Kaplan-Meier survival analysis will be used to compare the differences in overall survival between the two groups. The study aims to evaluate the application value of tumor organoid drug sensitivity experiments in guiding neoadjuvant chemotherapy for bladder cancer.

Research Objective: By observing the clinical efficacy of neoadjuvant chemotherapy guided by the tumor organoid drug sensitivity method in bladder cancer patients, this study aims to evaluate the application value of tumor organoid drug sensitivity experiments in guiding individualized neoadjuvant chemotherapy for bladder cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 18-80 years, any gender; 2. Patients with cT2~4aNxM0 MIBC who need neoadjuvant chemotherapy; 3. Patients who have not previously received systemic chemotherapy; 4. Patients who can tolerate platinum-based combination neoadjuvant chemotherapy; 5. ECOG performance status of 0-2; 6. According to the investigator's judgment, able to comply with the trial protocol, have good adherence, can cooperate in monitoring adverse events and efficacy, and participate in follow-up; 7. Voluntarily participate in this clinical trial, understand the study procedures, and have signed the informed consent form for participation.

Exclusion Criteria:

* 1. Patients with muscle-invasive bladder cancer (MIBC) with clinical stage T4b or distant metastasis, or the patient's physical condition is assessed to be intolerable to radical cystectomy; 2. Immunodeficiency or damage (such as AIDS patients, patients on immunosuppressants or radiotherapy); 3. Study participants who are known to be allergic or allergic to study drugs, similar drugs, excipients; 4. Those who have been taking hormonal drugs for a long time or have a history of drug abuse and dependence; 5. Those who have recently planned to become pregnant or are already pregnant or breastfeeding; 6. Abnormal blood routine, liver and kidney function and coagulation indicators: (1 or more can be considered abnormal)

  1) Neutrophil count (ANC) ≤1.5×109/L; 2) White blood cell count (WBC) ≤3.0×109/L; 3) Platelet count (PLT) ≤90×109/L; 4) Hemoglobin (HB) ≤90g/L; 5) Total bilirubin (TBIL) ≥1.5 × institutional upper limit of normal (ULN); 6) Estimated glomerular filtration rate (eGFR) ≤ 30 ml/min/1.73m²; 7) International normalized ratio (INR) and activated partial thromboplastin time (APTT) ≥ULN (except for patients receiving anticoagulant therapy, which need to be considered clinically acceptable by the investigator); 7. Study participants have other factors that could cause forced termination of this study, such as: 7) Patients have a previous or current diagnosis of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML); 8) Previous history of definite neurological or psychiatric disorders, including epilepsy or dementia; 9) Concomitant diseases that seriously endanger the safety of patients or affect the completion of the study (such as severe hypertension, diabetes, thyroid disease, etc.); 10) Other serious diseases require combined treatment, with serious laboratory abnormalities; 11) Other serious diseases accompanied by family or social factors that will affect the safety of research participants, or the collection of data and samples, etc.; 12) Have uncontrolled intercurrent illness, including but not limited to ongoing or active infection requiring treatment, symptomatic congestive heart failure, unstable angina pectoris, or arrhythmia; 8. Those who are not suitable to participate in this study in the opinion of the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients who need to come to the research center for treatment of bladder cancer
Sampling Method: Non-Probability Sample
Enrollment: 254 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
One-year OS ,Three-year OS and five-year OS | 2026.01.01-2030.12.31
  One-year overall survival rate, three-year overall survival rate, five-year overall survival rate

SECONDARY OUTCOMES:
One-year PFS ,Three-year PFS and five-year PFS | 2026.01.01-2030.12.31
  One-year progression-free survival rate, three-year progression-free survival rate, five-year progression-free survival rate.
CRR,CPR,ORR | 2025.01.01-2025.12.31
  Clinical complete remission rate, clinical partial remission rate, objective response rate

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong University, Jinan, China

IPD SHARING:
Plan to Share IPD: Yes